CLINICAL TRIAL: NCT01174888
Title: Phase I Study of the Combination of Midostaurin, Bortezomib, and Chemotherapy in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Phase I Combination of Midostaurin, Bortezomib, and Chemo in Relapsed/Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alison Walker (Other)
Collaborators: Novartis (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Alison Walker, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09111; NCI-2010-01335 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia With Multilineage Dysplasia Following; Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Congenital Abnormalities | interventions — midostaurin; Bortezomib; Mitoxantrone; Etoposide; Podophyllotoxin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP I (Dose levels 1-2): (Experimental): Patients receive midostaurin orally (PO) twice daily on days 1-14 and bortezomib intravenously (IV) on days 1, 4, 8, and 11. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: midostaurin; Drug: Bortezomib
- GROUP II (Dose levels 3-6) (Experimental): Patients receive mitoxantrone hydrochloride IV over 10 minutes, etoposide IV over 1 hour, and cytarabine IV over 6 hours on days 1-6. Patients also receive midostaurin PO twice daily on days 8-21 and bortezomib IV on days 8, 11, 15, and 18. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: midostaurin; Drug: Bortezomib; Drug: mitoxantrone hydrochloride; Drug: etoposide; Drug: cytarabine

INTERVENTIONS:
Drug: midostaurin — Drug midostaurin, Given orally given twice daily days 1-14
  Other Names: N-benzoyl-staurosporine; PKC412
Drug: Bortezomib — Bortezomib given IV on days 1, 4, 8, and 11
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: mitoxantrone hydrochloride — Patients receive mitoxantrone hydrochloride IV over 10 minutes
  Other Names: CL 232315; DHAD; DHAQ; dihydroxyanthracenedione; mitoxantrone HCl; Novantrone
  Arms: GROUP II (Dose levels 3-6)
Drug: etoposide — Patients receive etoposide IV over 1 hour
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; epipodophyllotoxin; VePesid; VP-16; VP-16-213
  Arms: GROUP II (Dose levels 3-6)
Drug: cytarabine — Patients receive cytarabine IV over 6 hours on days 1-6
  Other Names: ARA-C; ARA-cell; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
  Arms: GROUP II (Dose levels 3-6)

SUMMARY:
RATIONALE: Bortezomib and midostaurin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as mitoxantrone hydrochloride, etoposide, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib and midostaurin together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with midostaurin with or without combination chemotherapy in treating patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of bortezomib in combination with midostaurin and intensive chemotherapy in patients with relapsed/refractory acute myeloid leukemia (AML).

II. To define the specific toxicities and the dose limiting toxicity (DLT) of midostaurin and bortezomib in combination with intensive chemotherapy in relapsed/refractory AML.

SECONDARY OBJECTIVES:

I. To determine the rate of complete remission (CR) of midostaurin and bortezomib in combination with intensive chemotherapy. II. To determine the overall response rate (ORR). III. To characterize the biological activity of midostaurin and bortezomib to potentially increase endogenous phosphatase activity and therefore inhibit aberrant tyrosine kinases by assessing FLT3 and KIT tyrosine kinase activity as well as SHP-1(Anti-Src Homology Phosphatase-1)phosphatase activity. IV. To correlate the biological activity of midostaurin and bortezomib to potentially increase endogenous phosphatase activity with clinical response. V. To conduct pharmacokinetic studies of midostaurin and bortezomib together and in combination with intensive chemotherapy.

VI. To determine the efficacy of midostaurin and bortezomib in combination with intensive chemotherapy at the maximum tolerated dose in patients with FLT3 or KIT tyrosine kinase mutations.

OUTLINE:

This is a dose escalation study of bortezomib. Patients are assigned to 1 of 2 treatment groups. GROUP I (Dose levels 1-2): Patients receive oral midostaurin twice daily on days 1-14 and bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. GROUP II (Dose levels 3-6): Patients receive mitoxantrone hydrochloride IV over 10 minutes, etoposide IV over 1 hour, and cytarabine IV over 6 hours on days 1-6. Patients also receive oral midostaurin twice daily on days 8-21 and bortezomib IV on days 8, 11, 15, and 18. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria

* Patients age >18 with relapsed or refractory acute myeloid leukemia by WHO criteria are eligible for dose levels 1 and 2. Patients age >18 and ≤ 70 with relapsed or refractory acute myeloid leukemia by WHO criteria are eligible for dose levels 3 through 6. Patients with secondary AML are eligible
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* Patients must have adequate organ function as defined below:

  * total bilirubin <2.0mg/dL or ≤1.5 ULN(institutional upper limit of normal)
  * AST(aspartate aminotransferase)(SGOT)/ALT(Alanine aminotransferase) (SGPT) <2.5 X institutional ULN
  * creatinine <1.7 mg /dL
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. If the patient does not agree, the patient is not eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willingness to sign the written informed consent document
* Patients must have recovered from the toxicity of prior therapy to less than Grade 2
* Patients status post prior hematopoietic stem cell transplantation are eligible

Exclusion criteria

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Hydroxyurea may be administered until initiation of treatment on the study
* Patients receiving any other investigational agents or patients that have received other investigational agents within 14 days of enrollment
* Patients with active central nervous system disease or with granulocytic sarcoma as sole site of disease
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to midostaurin, bortezomib, mitoxantrone, etoposide or cytarabine that are not easily managed. Patient has a hypersensitivity to bortezomib, boron, or mannitol.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, uncontrolled hypertension, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Ejection fraction <50%
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Pregnant women or women who are breastfeeding are excluded from this study.
* Patients with pre-existing Grade 2 or higher neuropathy or other serious neurologic toxicity that would significantly increase risk of complications from bortezomib therapy are excluded.
* Patients with a known confirmed diagnosis of HIV infection (due to concern for increased toxicity with the regimen in combination with HAART) or active viral hepatitis.
* Patients with any pulmonary infiltrate including those suspected to be of infectious origin. In particular, patients with resolution of clinical symptoms of pulmonary infection but with residual pulmonary infiltrates on chest x-ray are not eligible until pulmonary infiltrates have completely resolved.
* Patients who have had any surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) within 14 days of Day 1.
* Patients with advanced malignant solid tumors are excluded.
* Patients with known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of midostaurin.
* Patients with prior midostaurin treatment are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) of bortezomib and midostaurin in combination with MEC salvage chemotherapy | up to 28 months
  Maximum tolerated dose of bortezomib and midostaurin in combination with MEC(mitoxantrone, etoposide,cytarabine)salvage chemotherapy. Specific toxicities and Dose-limiting toxicity of midostaurin and bortezomib in combination with intensive chemotherapy in relapsed/refractory AML.

SECONDARY OUTCOMES:
determine the rate of complete remission (CR) | up to 28 months
  To determine the rate of complete remission (CR) of midostaurin and bortezomib in combination with intensive chemotherapy.
Determine the overall response rate (ORR) | up to 28 months
  To determine the overall response rate (ORR)
Characterize the biological activity of midostaurin and bortezomib | up to 28 months
  Characterize the biological activity of midostaurin and bortezomib to potentially increase endogenous phosphatase activity and therefore inhibit aberrant tyrosine kinases by assessing FLT3(fetal liver kinase-2)and KIT tyrosine kinase activity as well as SHP-1 phosphatase activity.
Correlate the biological activity of midostaurin and bortezomib | up to 28 months
  To correlate the biological activity of midostaurin and bortezomib to potentially increase endogenous phosphatase activity with clinical response.
Conduct pharmacokinetic studies of midostaurin and bortezomib | up to 28 months
  To conduct pharmacokinetic studies of midostaurin and bortezomib together and in combination with intensive chemotherapy.
Determine the efficacy of midostaurin and bortezomib | up to 28 months
  To determine the efficacy of midostaurin and bortezomib in combination with intensive chemotherapy at the maximum tolerated dose in patients with FLT3 or KIT tyrosine kinase mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Walker, MD, Principal Investigator — The Ohio State University James Cancer Hospital
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Walker AR, Wang H, Walsh K, Bhatnagar B, Vasu S, Garzon R, Canning R, Geyer S, Wu YZ, Devine SM, Klisovic R, Blum W, Marcucci G. Midostaurin, bortezomib and MEC in relapsed/refractory acute myeloid leukemia. Leuk Lymphoma. 2016 Sep;57(9):2100-8. doi: 10.3109/10428194.2015.1135435. Epub 2016 Jan 19. PMID 26784138
- See also: Jamesline — http://cancer.osu.edu